CLINICAL TRIAL: NCT04908020
Title: Coping and Post Traumatic Stress Disorder in Children and Adolescents During Cancer Follow-up Care: a Prospective Observational Cohort Study
Brief Title: Coping and Post Traumatic Distress in Children and Adolescents During Cancer Follow-up Care
Status: Completed | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Rosanna Martin, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: FOLLOWUP_PTSD
Record Dates: First submitted 2021-02-10; First posted 2021-06-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Cancer; Follow-up Care
Keywords: post-traumatic stress; coping; pediatric cancer; follow-up
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Follow up: The group is made up by children and adolescents, aged from 9 to 17, who received a cancer diagnosis, who completed oncological treatment and who are included in a clinical follow-up program since less than 3 years.
  Furthermore, the study involves one parent for each patient to collect demographics and clinical data.
  Interventions: Other: Follow-up patients

INTERVENTIONS:
Other: Follow-up patients — The intervention consists in the assessment of some psychological aspects (post traumatic stress symptoms and coping) of cancer patients in follow-up care, through specific tests. Each patient fills out the test battery during the psychological consult. At the same time, it is involved a parent to collect personal and clinical data through an ad hoc questionnaire.

SUMMARY:
To explore the presence of post traumatic disorder and its association with coping strategies in children and adolescents during cancer follow-up care.

Hypothesis: the investigators expect a reduction of post traumatic symptoms according to adequate coping strategies (eg. approach coping styles).

DETAILED DESCRIPTION:
Oncological disease in childhood or adolescence can represent a highly traumatic experience, considering its physical, psychological and social consequences in the short and long term. The literature has investigated this population both in the acute phase of the disease and at the end of the therapies to explore the potentially traumatic effects of this experience. While some studies support the non-incidence of post-traumatic symptoms related to the disease and underline a post-traumatic growth, other studies confirm a high risk of developing post-traumatic symptoms. This risk increases according to specific demographic (eg. age of diagnosis) and clinical (eg. type of disease, of treatments, etc.) characteristics. The literature also points out that these consequences can be mediated by some factors, including coping strategies, that is the way patients manage stress.

The study aims: to investigate the presence of post-traumatic symptoms in patients out of therapy and in follow-up care; to explore the possible association between this post-traumatic symptomatology and the coping strategies used by the patients; to focus the possible correlation between post traumatic symptoms, coping and the demographic and clinical characteristics of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in cancer follow-up care since less than 3 years
* Scheduled to follow-up appointement
* Italian speaking
* Patients' and parents' consent

Exclusion Criteria:

- Cognitive and/or developmental impairment

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population is made up by children and adolescents, aged from 9 to 17, who received a cancer diagnosis, who completed oncological treatment and who are "out of therapies". Furthermore, they have to be included in a clinical follow-up program since less than 3 years.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
post traumatic stress symptoms | Post-traumatic Stress Symptoms are assessed at the first psychological consult since beginning of the study, indipendently from follow up time. Is a single assessment for every partecipant.
  Trauma Symptom Checklist for Children (TSCC-A) is a self report questionnaire that assess children and adolscents' post-traumatic symptoms with 5 clinical scales: anxiety, depression, anger, post-traumatic distress, dissociation (the complete version TSCC includes sexual interest scale). It can be filled out by children and adolescents aged from 8 to 17. Each patient has to read a list of thoughts, feelings and behaviors and to rate their frequency on a 4-point Likert scale (1= never; 5= always).
coping strategies type_12-17 | Coping strategies are assessed at the first psychological consult since beginning of the study, indipendently from follow up time. Is a single assessment for every partecipant.
  Coping Responsing Inventory (youth version; CRI-YOUTH): self report questionnaire that identify and monitor adolescents' coping strategies to manage stress. The CRI-youth assess coping strategies of youth, aged from 12 to 18, using 8 scales: these scales cover the areas of approach coping styles (Logical Analysis, Positive Reappraisal, Seeking Guidance and Support, and Problem Solving) and avoidant coping styles (Cognitive Avoidance, Acceptance or Resignation, Seeking Alternative Rewards, and Emotional Discharge).
  CRI-YOUTH is rated on a 4-point Likert scale (1= never; 5= always), with T-points from 20 to 80+ with higher scores indicating a higher usage of a coping strategy.
  Each patient had to read a list of sentences about the cognitive and behavioral responses to cope with a stressful situation and to rate their use on a 4-point Likert scale (1= never; 5= always).
coping strategies type_9-11 | Coping strategies are assessed at the first psychological consult since beginning of the study, indipendently from follow up time. Is a single assessment for every partecipant.
  Children's Coping Strategies Checklist-Revision1 (CCSC-R1) is a self report questionnaire that identify children's coping strategies to manage stress. It contains 54 items organized in 13 subscales, loading five dimensions: problem-focused coping and positive cognitive restructuring, distraction coping strategies, avoidance coping strategies, and support-seeking strategies. Both problem-focused coping and positive cognitive restructuring are considered dimensions of active coping. Children request to assess how frequently they usually adopt the coping strategies described in the item on a 4-point Likert scale (1= never; 5= always).For each scale and subscale, the score is the mean of scores of the scale items.

SECONDARY OUTCOMES:
demographic data | Both patients and parents fill out the ad-hoc questionnaire at the first psychological consult since beginning of the study, indipendently from follow up time. Is a single assessment for every partecipant.
  The questionnaire includes a section devoted to demographics (i.e., gender, present age, age at the time of diagnosis, nationality, etc.) and to clinical data (eg. type of disease, treatments, other traumatic events, etc.). Only the parents' version contains the section related to personal and clinical data. An additional section aims to explore the thoughts, feelings and behaviour of child, adolescents and parents in the main moments of the patient's disease (communication of diagnosis, treatment, follow-up) through open and closed questions.
  Data are qualitative, no scoring, and will be helpful for cathegorization during statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Stagi, MD, Study Director — Meyer Children's Hospital IRCCS; Rosanna Martin, MSc, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Children's Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Decision has to be shared with the Clinical Trial Office of the Hospital

REFERENCES:
- [Background] Bremner JD. Acute and chronic responses to psychological trauma: where do we go from here? Am J Psychiatry. 1999 Mar;156(3):349-51. doi: 10.1176/ajp.156.3.349. No abstract available. PMID 10080546
- [Background] Briere J, Kaltman S, Green BL. Accumulated childhood trauma and symptom complexity. J Trauma Stress. 2008 Apr;21(2):223-6. doi: 10.1002/jts.20317. PMID 18404627
- [Background] Cloitre M, Stolbach BC, Herman JL, van der Kolk B, Pynoos R, Wang J, Petkova E. A developmental approach to complex PTSD: childhood and adult cumulative trauma as predictors of symptom complexity. J Trauma Stress. 2009 Oct;22(5):399-408. doi: 10.1002/jts.20444. Epub 2009 Sep 30. PMID 19795402
- [Background] Compas BE, Connor-Smith JK, Saltzman H, Thomsen AH, Wadsworth ME. Coping with stress during childhood and adolescence: problems, progress, and potential in theory and research. Psychol Bull. 2001 Jan;127(1):87-127. PMID 11271757
- [Background] Duran B. Posttraumatic growth as experienced by childhood cancer survivors and their families: a narrative synthesis of qualitative and quantitative research. J Pediatr Oncol Nurs. 2013 Jul-Aug;30(4):179-97. doi: 10.1177/1043454213487433. Epub 2013 May 8. PMID 23657991
- [Background] Kangas M. DSM-5 Trauma and Stress-Related Disorders: Implications for Screening for Cancer-Related Stress. Front Psychiatry. 2013 Oct 2;4:122. doi: 10.3389/fpsyt.2013.00122. No abstract available. PMID 24106482
- [Background] Koutna V, Jelinek M, Blatny M, Kepak T. Predictors of Posttraumatic Stress and Posttraumatic Growth in Childhood Cancer Survivors. Cancers (Basel). 2017 Mar 16;9(3):26. doi: 10.3390/cancers9030026. PMID 28300764
- [Background] Billings AG, Moos RH. The role of coping responses and social resources in attenuating the stress of life events. J Behav Med. 1981 Jun;4(2):139-57. doi: 10.1007/BF00844267. PMID 7321033
- [Background] Phipps S, Long A, Hudson M, Rai SN. Symptoms of post-traumatic stress in children with cancer and their parents: effects of informant and time from diagnosis. Pediatr Blood Cancer. 2005 Dec;45(7):952-9. doi: 10.1002/pbc.20373. PMID 15806541
- [Background] Phipps S, Steele R. Repressive adaptive style in children with chronic illness. Psychosom Med. 2002 Jan-Feb;64(1):34-42. doi: 10.1097/00006842-200201000-00006. PMID 11818584
- [Background] Scrignaro M, Barni S, Magrin ME. The combined contribution of social support and coping strategies in predicting post-traumatic growth: a longitudinal study on cancer patients. Psychooncology. 2011 Aug;20(8):823-31. doi: 10.1002/pon.1782. Epub 2010 Jun 3. PMID 20878872
- [Background] Sposito AM, Silva-Rodrigues FM, Sparapani Vde C, Pfeifer LI, de Lima RA, Nascimento LC. Coping strategies used by hospitalized children with cancer undergoing chemotherapy. J Nurs Scholarsh. 2015 Mar;47(2):143-51. doi: 10.1111/jnu.12126. Epub 2015 Jan 31. PMID 25639151
- [Background] Tremolada M, Bonichini S, Basso G, Pillon M. Post-traumatic Stress Symptoms and Post-traumatic Growth in 223 Childhood Cancer Survivors: Predictive Risk Factors. Front Psychol. 2016 Feb 29;7:287. doi: 10.3389/fpsyg.2016.00287. eCollection 2016. PMID 26973578
- [Background] Zeltzer LK, Recklitis C, Buchbinder D, Zebrack B, Casillas J, Tsao JC, Lu Q, Krull K. Psychological status in childhood cancer survivors: a report from the Childhood Cancer Survivor Study. J Clin Oncol. 2009 May 10;27(14):2396-404. doi: 10.1200/JCO.2008.21.1433. Epub 2009 Mar 2. PMID 19255309